CLINICAL TRIAL: NCT04893902
Title: An Innovative Approach for Auricular Rehabilitation Using Two Types Digital Impression Versus Conventional Techniques:
Brief Title: Digital VS. Conventional Ear Impression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Mahmoud Dohiem (Other Government)
Responsible Party: Sponsor-Investigator, Mohamed Mahmoud Dohiem, lecture prosthetic department zagazig university egypt, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dohiem md
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Patient Loss His Ear and Need Auricular Prosthesis
Keywords: Ear impression -Ear scanning-intraoral scanner-scannin marker-ear prosthesis

STUDY DESIGN:
Intervention Model Description: control clinical rial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional ear impression (Active Comparator)
  Interventions: Device: medit intra oral scanner
- digital auricular impression without marker using intra oral scanner (Experimental)
  Interventions: Device: medit intra oral scanner
- digital auricular impression with marker using intra oral scanner (Experimental)
  Interventions: Device: medit intra oral scanner

INTERVENTIONS:
Device: medit intra oral scanner — ear scanning with intra oral scanner

SUMMARY:
What is known:

Ear impressions are made in conventional manner by impression materials which may affect the accuracy of the obtained data and consume time and effort .

What this study adds:

Predesigned ear markers facilitate ear scanning using an intraoral scanner that decreases the probability of in-accuracies using the conventional manner with less time and effort

DETAILED DESCRIPTION:
Prosthodontic maxillofacial rehabilitation of acquired or congenital ear defects is considered a challenging procedure. This clinical trial introduces a novel approach for digital scanning of the unaffected contralateral ear using an intraoral scanner in comparison to the conventional impression techniques. CAD/CAM is a very promising design and fabrication of an auricular prosthesis for patients with unilateral ear defects.

Purpose: This study aims to compare digital impression technique using an intra-oral digital scanner IOSfor the unaffected ear with markers /without markers versus traditional techniques with hydro colloidal impression materials.

ELIGIBILITY:
Inclusion Criteria:

* any normal patient

Exclusion criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2021-05-16 (Estimated); Study Completion 2021-05-17 (Estimated)

PRIMARY OUTCOMES:
total deviation between Conventional auricular impression and two types of digital impression | 1 day

SECONDARY OUTCOMES:
total deviation between two types of digital impression | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud dohiem, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dohiem MM, Emam NS, Abdallah MF, Abdelaziz MS. Accuracy of digital auricular impression using intraoral scanner versus conventional impression technique for ear rehabilitation: A controlled clinical trial. J Plast Reconstr Aesthet Surg. 2022 Nov;75(11):4254-4263. doi: 10.1016/j.bjps.2022.08.002. Epub 2022 Aug 5. PMID 36117136